CLINICAL TRIAL: NCT05703568
Title: Effect of the Group-based Virtual Reality Training on Activities of Daily Living in Elderly: a Randomized Controlled Trial
Brief Title: Effect of the Virtual Reality Training in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Oznur Fidan, Principal investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gazi University
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-07

CONDITIONS: Elderly

STUDY DESIGN:
Intervention Model Description: Each participant will be requested to draw either number one, number two or number three from a box. Number one will be allocated to group 1, number two will be allocated o group 2 and number two will be allocated o group 3. The group 1 consists of 14 elderly participants who received intervention protocol of group- based virtual reality training program in which total 16-sessions were given for twice a week for eight weeks for 45-minutes. The group 2 consists of 14 elderly participants who received intervention protocol of individual virtual reality training in which total 16-sessions were given for twice a week for eight weeks for 45-minutes. The group 3 consists of 14 elderly participants will continue their routine daily activities.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group- based virtual reality training (Experimental): Individuals in this arm will be received intervention protocol of group- based virtual reality training program in which total 16-sessions were given for twice a week for eight weeks for 45-minutes.
  Interventions: Other: virtual reality
- Individual virtual reality training (Experimental): Individuals in this arm will be received intervention protocol of individual virtual reality training program in which total 16-sessions were given for twice a week for eight weeks for 45-minutes.
  Interventions: Other: Virtual reality
- Control group (No Intervention): Individuals in this arm will continue their routine daily activities.

INTERVENTIONS:
Other: virtual reality — 14 elderly participants receive intervention protocol of group- based virtual reality training program (XBOX Kinect games: Your Shape: Fitness Evolved) in which total 16-sessions were given for twice a week for eight weeks for 45-minutes.
  Arms: Group- based virtual reality training
Other: Virtual reality — 14 elderly participants receive intervention protocol of individual virtual reality training program (XBOX Kinect games: Your Shape: Fitness Evolved) in which total 16-sessions were given for twice a week for eight weeks for 45-minutes.
  Arms: Individual virtual reality training

SUMMARY:
The study aims to investigate the efficacy of group-based exercises using virtual reality on activities of daily living in elderly population.

DETAILED DESCRIPTION:
As a result of morphological and functional changes that occur with aging, complications such as decrease in muscle mass, flexibility and muscle strength, decrease in sleep quality, social isolation and chronic diseases develop and cause a decrease in independence in activities of daily living (ADL). Increasing physical activity in the elderly is effective in maintaining general health status and maintaining independence during activities of daily living (ADL). However, the level of the participation to physical activities is quite low in old age. It's known that group-based exercises and technology-supported exercise training with virtual reality games increase participation in physical activity and improve motor functions and ADL. But, there is no study examining the effect of technology-supported group exercises on ADLs in the elderly. Therefore, the aim of our study is to find out the effects of technology-supported group exercises on ADLs in the elderly over 65 years of age.

The forty-two participants will be recruited and divided into three equal groups randomly. The group 1(n=14) will perform group-based virtual reality training and group 2(n=14) will receive individual virtual reality training for 45-minutes, twice a week for eight weeks. The third group group 3(n=14) will determined as the control group and they will continue their routine daily activities. Primary outcome measure will be Barthel Index of Activities of Daily Living. Secondary outcome measures will be Physical Activity Scale for the Elderly (PASE), Timed Up and Go (TUG) test, Single Leg Stance Test (SLST), Six Minute Walk Test, Geriatric Depression Scale (GDS), Physical Activity Enjoyment Scale (Paces).

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 65 age or older
* can ambulate independently

Exclusion Criteria:

* elderly individuals who are suffering from any acute or unstable illness or medical condition
* elderly individuals who are unable to understand the treatment protocol.
* elderly individuals who are suffering from any kind of visual, auditory and neural or vestibular system disorders.
* History of surgery in the last 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Barthel Index for Activities of Daily Living | 8 weeks
  The Barthel Index, measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Total scores range from 0 - 20, with lower scores indicating increased disability.

SECONDARY OUTCOMES:
Physical Activity Scale for the Elderly | 8 weeks
  Physical Activity Scale for the Elderly is a brief (5 minutes) and easily scored survey designed specifically to assess physical activity in epidemiological studies of person age 65 years and older. The total score ranges from 0 to 400 or more and high scores show better physical activity levels.
Timed Up and Go (TUG) | 8 weeks
  Time Up and Go is a very simple, quick, valid, reliable and an objective test which is used for the assessment of balance and mobility.
Single Leg Stance Test (SLST) | 8 weeks
  Single Leg Stance Test (SLST) test is used to assess balance. For the test, volunteers were asked to lift one foot without touching the support leg.
Six minute walk test | 8 weeks
  Six minute walk test is used to assessment of walking related performance fatigability
Geriatric Depression Scale | 8 weeks
  This instrument evaluate depressive symptoms using yes/no answers. Of the 15 items, 10 indicate the presence of depression when answered positively while the other 5 are indicative of depression when answered negatively
Physical Activity Enjoyment Scale (Paces) | 8 weeks
  This scale measures enjoyment during physical activity through with 5 items from the original18 items.
Mini Mental State Test | Baseline
  Mini Mental State Test,30-point test, will be used for cognitive assessment.A score of 23 or lower is indicative of cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided